CLINICAL TRIAL: NCT05977114
Title: 4Rs for a Better Family (Review, Refresh, Restore, Rebuild) 家好之四重計劃: 重溫、重整、重塑、重建
Brief Title: 4Rs for a Better Family
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Nancy Xiaonan Yu, Associate Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4Rs for a Better Family
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Family Relations

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4Rs Group (Experimental)
  Interventions: Behavioral: family conflict intervention group
- 4As Group (Active Comparator)
  Interventions: Behavioral: handicraft-making group

INTERVENTIONS:
Behavioral: family conflict intervention group — The family conflict preventive intervention includes the introduction to the occurrence of family conflicts, communication skills training, and role play to practice the skills.
  Arms: 4Rs Group
Behavioral: handicraft-making group — The group involves handicraft-making.
  Arms: 4As Group

SUMMARY:
The goal of this clinical trial is to learn about the effects of a family conflict intervention in Chinese New Arrival families in Hong Kong.

The main questions it aims to answer are:

* Is the family conflict intervention group more effective to improve adaptive parent-child conflict resolution skills compared to the control group?
* Is the family conflict intervention group more effective to reduce parent-child conflicts compared to the control group?
* Is the family conflict intervention group more effective to improve adaptive parental conflict resolution skills compared to the control group?
* Is the family conflict intervention group more effective to enhance family harmony compared to the control group?
* Is the family conflict intervention group more effective to enhance family resilience compared to the control group?

Participants will be randomly assigned to one of the two groups: the family conflict intervention group and the handcraft-making group. For each group, parents will participate in 3 sessions independently, children will participate in 2 sessions independently, and parents and children will jointly participate in 1 session. Each session takes around 2 hours, and it takes 4 weeks to complete the full intervention. The family conflict intervention sessions include an introduction to the occurrence of family conflicts, communication skills training to prevent and address conflicts, and role play to practice the skills, etc.

Researchers will compare the family conflict intervention group and the handcraft-making group to see if the family conflict intervention group is effective in promoting conflict resolution skills, reducing family conflicts, and enhancing family resilience.

ELIGIBILITY:
Inclusion Criteria:

1. Parents who have newly arrived in Hong Kong for less than seven years, and their children who are studying in primary school grade 4 to secondary school form 3; or
2. New arrivals who have settled in Hong Kong for less than seven years and are studying in primary school grade 4 to secondary school form 3, and their parents; and
3. Parents and children must live together; and
4. Parents and children must participate together

Exclusion Criteria:

1. Self-reported serious emotional or mental illness by parent or child, or
2. Children with special learning needs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Parent-child conflicts | Baseline, 4 weeks, 8 weeks
  Parent-child conflicts are measured by the frequency and intensity of parent-child conflicts (Yau & Smetana, 1996). Possible scores for conflict frequency range from 0 (not at all) to 4 (4 times or above). A higher score indicates a higher level of parent-child conflict frequency. Possible scores for conflict intensity range from 1 (none) to 5 (severe). A higher score indicates more severe parent-child conflicts.
Parent-child conflict resolution | Baseline, 4 weeks, 8 weeks
  Parent-child conflict adaptive resolution strategy is measured by the subscale of the Parent-Child Conflict Response Strategy Scale (Sun, 2019). The four items are each rated on a five-point scale, which is from 1 (never) to 5 (always). A higher score indicates a higher level of adaptive parent-child conflict resolution.
The Chinese version of the Rahim Organizational Conflict Inventory-II | Baseline, 4 weeks, 8 weeks
  Couple conflict and problem-solving will be measured by the subscale of the Chinese version of the Rahim Organizational Conflict Inventory-II (ROC-II; Rahim, 1983; Chang & Lu, 2007). The subscale includes 7 items. Each item is rated on a five-point scale. A higher score indicates a higher level of adaptive couple conflict resolution.
Family Harmony Scale | Baseline, 4 weeks, 8 weeks
  Family Harmony will be measured by the Family Harmony Scale (Fabrizio et al., 2015). The scale includes 8 items. Each item is rated on a five-point scale. A higher score indicates a higher level of family harmony.
Family Resilience Quetionnaire | Baseline, 4 weeks, 8 weeks
  Family Resilience will be measured by the Walsh Family Resilience Questionnaire (Walsh, 2015). We selected 9 representative questions from the original questionnaire for our study. Each item is rated on a five-point scale. A higher score indicates a higher level of family resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Nancy YU, Doctoral, Principal Investigator — City University of Hong Kong
Locations (1):
- International Social Service Hong Kong Branch, Hong Kong, China